CLINICAL TRIAL: NCT04174378
Title: A Comparison Of Progestogens Plus GnRH Agonist Versus Progestogens Only In Luteal Phase Support In IVF Women: A Retrospective Single Centre Experience
Brief Title: Luteal Phase Support In IVF Women Using GnRH Agonist
Status: Completed | Type: Observational
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Azrai Abu, Principal Investigator, National University of Malaysia
Other Study IDs: PPI/111/8/JEP-2018-619
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: IVF; Luteal Phase Defect
Keywords: Luteal phase support; GnRH agonist; in vitro fertilization
MeSH Terms: interventions — Triptorelin Pamoate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GnRH agonist with progestogen support
  Interventions: Drug: Decapeptyl 0.2mg
- progestogen support only

INTERVENTIONS:
Drug: Decapeptyl 0.2mg — IM Decapeptyl o.2 mg was given 2 days before embryo transfer
  Groups: GnRH agonist with progestogen support

SUMMARY:
Lately, the role of GnRH agonist as luteal phase support has been recommended by various studies though the mechanism is still debatable. It has been postulated that GnRH agonist might support the corpus luteum by stimulating the secretion of luteinizing hormone by pituitary gonadotroph cells, or by acting directly on the endometrium through the locally expressed receptors.

Therefore, this study was designed to evaluate effects of the additional of single-dose GnRH agonist to the routine progestogens use for luteal phase support on IVF outcome as compared to progestogens only. The biochemical pregnancy rates, clinical pregnancy rates, live birth rates and miscarriage rate between these regimes were compared. The hypothesis of this study was women with addition of GnRH agonist as luteal phase support have higher biochemical pregnancy rate, clinical pregnancy rate and live birth rate compare to patient with progestogens only luteal phase support.

DETAILED DESCRIPTION:
This was a retrospective study on selected patients who underwent IVF treatment under MAC (Medically Assisted Conception) Unit, University Kebangsaan Malaysia Medical Centre for the period of June 2015-June 2018. Their medical records were reviewed, and data analysed.

The sample size was calculated using Power & Sample Size Calculator by Dupont & Plummer 1998 for dichotomous response version 3.1.2 [6]. Based on this formula, a is the type I error probability for a two-sided test allowable about 5% in this study. The power of certainty is the percentage of estimated power of this study. On the other hand, p0 is the probability of the outcome for GnRH agonist used as luteal phase support by Zafardoust et al. [7] which is 30% (0.30). The p1 is the probability of the outcome in an experimental subject which expected in this study based on similar objective of higher rate of implantation with GnRH agonist. The investigators set the p1 is 0.50 as overall literature suggest that at cumulative successful of implantation post GnRH is around 30-50%. The m is the ratio of control to experimental subjects which is 1 to 1 in this study. Generated sample size from this program is 93 for one arm which result in total sample size is 186. The investigators then added 10% of additional sample for any bias or loss of data during follow up which concluded total sample size to be at least 200 samples (100 patients each arm).

All women who underwent control-ovarian stimulation (COH) regime using either gonadotrophin combination with GnRH antagonist protocol or mild stimulation protocol using oral letrozole or clomiphene citrate were included in this study. All women underwent follicle tracking by transvaginal ultrasound until dominant follicle size reached (>18mm). IM Ovitrelle (6500 IU) was given and proceed with oocyte retrieval (OR) at least 35-36 hours under transvaginal ultrasonography guidance. The 17-gauge single -lumen needles used for oocyte retrieval under sedation.

ICSI were performed according to local protocol. Zygotes were cultured up to day 5 in G1 medium (Vitrolife). On day 5, embryos were graded according to previously described criteria. One or two embryos were transferred, depending on the morphological score and the developmental stage of the embryo, as well as the age of the patient.

Regardless the ovarian stimulation protocols, these women were assigned into two group; progestogens with additions of GnRH agonist and progestogen only for luteal phase support. Both groups were given routine progestogen support for two weeks duration started from the day of embryo transfer. This includes oral progestogen (Tablet Duphaston 10mg tds), vaginal progestogen (vaginal utrogestan 400mg bd) or intramuscular (IM Proluton 250 mg weekly) as prescribed by attending clinician .

In the first group, there were additional GnRH agonist administrated as a single dose of 0.2 mg decapeptyl given at day 3 after ICSI. The other group with no GnRH agonist given was the control group.

ELIGIBILITY:
Inclusion Criteria:

* underwent ICSI
* given progestogens plus GnRH agonist or progestogens only as luteal phase support.

Exclusion Criteria:

* different luteal phase support
* frozen embryo transfer and
* missing medical records data

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Data women underwent IVF treatment under MAC (Medically Assisted Conception) Unit, University Kebangsaan Malaysia Medical Centre for the period of June 2015-June 2018 were reviewed.
Sampling Method: Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Biochemical pregnancy rate | 14 days after embryo transfer
  serum B-HCG more than 5 mIU/ml
clinical pregnancy rate | 4 weeks after embryo transfer
  presence of gestational sac
live birth rate | beyond 24 weeks of gestation
  gestation more than 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Azrai Abu, Medical Degree, Principal Investigator — Department of Obstetrics and Gynecology, UKM Medical Centre
Locations (1):
- Medically Assisted Conception Unit, UKM Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beckers NG, Macklon NS, Eijkemans MJ, Ludwig M, Felberbaum RE, Diedrich K, Bustion S, Loumaye E, Fauser BC. Nonsupplemented luteal phase characteristics after the administration of recombinant human chorionic gonadotropin, recombinant luteinizing hormone, or gonadotropin-releasing hormone (GnRH) agonist to induce final oocyte maturation in in vitro fertilization patients after ovarian stimulation with recombinant follicle-stimulating hormone and GnRH antagonist cotreatment. J Clin Endocrinol Metab. 2003 Sep;88(9):4186-92. doi: 10.1210/jc.2002-021953. PMID 12970285
- [Result] Kolibianakis EM, Bourgain C, Platteau P, Albano C, Van Steirteghem AC, Devroey P. Abnormal endometrial development occurs during the luteal phase of nonsupplemented donor cycles treated with recombinant follicle-stimulating hormone and gonadotropin-releasing hormone antagonists. Fertil Steril. 2003 Aug;80(2):464-6. doi: 10.1016/s0015-0282(03)00663-0. No abstract available. PMID 12909519
- [Result] Smitz J, Bourgain C, Van Waesberghe L, Camus M, Devroey P, Van Steirteghem AC. A prospective randomized study on oestradiol valerate supplementation in addition to intravaginal micronized progesterone in buserelin and HMG induced superovulation. Hum Reprod. 1993 Jan;8(1):40-5. doi: 10.1093/oxfordjournals.humrep.a137871. PMID 8458924
- [Result] Pritts EA, Atwood AK. Luteal phase support in infertility treatment: a meta-analysis of the randomized trials. Hum Reprod. 2002 Sep;17(9):2287-99. doi: 10.1093/humrep/17.9.2287. PMID 12202415
- [Result] Tesarik J, Hazout A, Mendoza-Tesarik R, Mendoza N, Mendoza C. Beneficial effect of luteal-phase GnRH agonist administration on embryo implantation after ICSI in both GnRH agonist- and antagonist-treated ovarian stimulation cycles. Hum Reprod. 2006 Oct;21(10):2572-9. doi: 10.1093/humrep/del173. Epub 2006 Aug 22. PMID 16926261
- [Result] Dupont WD, Plummer WD Jr. Power and sample size calculations. A review and computer program. Control Clin Trials. 1990 Apr;11(2):116-28. doi: 10.1016/0197-2456(90)90005-m. PMID 2161310
- [Result] Zafardoust S, Jeddi-Tehrani M, Akhondi MM, Sadeghi MR, Kamali K, Mokhtar S, Badehnoosh B, Arjmand-Teymouri F, Fatemi F, Mohammadzadeh A. Effect of Administration of Single Dose GnRH Agonist in Luteal Phase on Outcome of ICSI-ET Cycles in Women with Previous History of IVF/ICSI Failure: A Randomized Controlled Trial. J Reprod Infertil. 2015 Apr-Jun;16(2):96-101. PMID 25927026
- [Result] Yildiz GA, Sukur YE, Ates C, Aytac R. The addition of gonadotrophin releasing hormone agonist to routine luteal phase support in intracytoplasmic sperm injection and embryo transfer cycles: a randomized clinical trial. Eur J Obstet Gynecol Reprod Biol. 2014 Nov;182:66-70. doi: 10.1016/j.ejogrb.2014.08.026. Epub 2014 Aug 27. PMID 25238659
- [Result] Qublan H, Amarin Z, Al-Qudah M, Diab F, Nawasreh M, Malkawi S, Balawneh M. Luteal phase support with GnRH-a improves implantation and pregnancy rates in IVF cycles with endometrium of <or=7 mm on day of egg retrieval. Hum Fertil (Camb). 2008 Mar;11(1):43-7. doi: 10.1080/14647270701704768. PMID 18320439
- [Result] Razieh DF, Maryam AR, Nasim T. Beneficial effect of luteal-phase gonadotropin-releasing hormone agonist administration on implantation rate after intracytoplasmic sperm injection. Taiwan J Obstet Gynecol. 2009 Sep;48(3):245-8. doi: 10.1016/S1028-4559(09)60297-7. PMID 19797013
- [Result] Ata B, Urman B. Single dose GnRH agonist administration in the luteal phase of assisted reproduction cycles: is the effect dependent on the type of GnRH analogue used for pituitary suppression? Reprod Biomed Online. 2010 Jan;20(1):165-6; author reply 167. doi: 10.1016/j.rbmo.2009.10.022. Epub 2009 Nov 10. No abstract available. PMID 20159003
- [Result] Ata B, Yakin K, Balaban B, Urman B. GnRH agonist protocol administration in the luteal phase in ICSI-ET cycles stimulated with the long GnRH agonist protocol: a randomized, controlled double blind study. Hum Reprod. 2008 Mar;23(3):668-73. doi: 10.1093/humrep/dem421. Epub 2008 Jan 12. PMID 18192671
- [Result] Kung HF, Chen MJ, Guua HF, Chen YF, Yi YC, Yen-Ping Ho J, Chou MM. Luteal phase support with decapeptyl improves pregnancy outcomes in intracytoplasmic sperm injection with higher basal follicle-stimulating hormone or lower mature oocytes. J Chin Med Assoc. 2014 Oct;77(10):524-30. doi: 10.1016/j.jcma.2014.07.001. Epub 2014 Aug 24. PMID 25160805
- [Result] Tesarik J, Hazout A, Mendoza C. Enhancement of embryo developmental potential by a single administration of GnRH agonist at the time of implantation. Hum Reprod. 2004 May;19(5):1176-80. doi: 10.1093/humrep/deh235. Epub 2004 Apr 7. PMID 15070873
- [Result] Davar R, Farid Mojtahedi M, Miraj S. Effects of single dose GnRH agonist as luteal support on pregnancy outcome in frozen-thawed embryo transfer cycles: an RCT. Iran J Reprod Med. 2015 Aug;13(8):483-8. PMID 26568750
- [Result] Benmachiche A, Benbouhedja S, Zoghmar A, Boularak A, Humaidan P. Impact of Mid-Luteal Phase GnRH Agonist Administration on Reproductive Outcomes in GnRH Agonist-Triggered Cycles: A Randomized Controlled Trial. Front Endocrinol (Lausanne). 2017 Jun 15;8:124. doi: 10.3389/fendo.2017.00124. eCollection 2017. PMID 28663739
- [Result] Pirard C, Donnez J, Loumaye E. GnRH agonist as novel luteal support: results of a randomized, parallel group, feasibility study using intranasal administration of buserelin. Hum Reprod. 2005 Jul;20(7):1798-804. doi: 10.1093/humrep/deh830. Epub 2005 May 12. PMID 15890740
- [Result] Pirard C, Donnez J, Loumaye E. GnRH agonist as luteal phase support in assisted reproduction technique cycles: results of a pilot study. Hum Reprod. 2006 Jul;21(7):1894-900. doi: 10.1093/humrep/del072. Epub 2006 Mar 23. PMID 16556673
- [Result] Fujii S, Sato S, Fukui A, Kimura H, Kasai G, Saito Y. Continuous administration of gonadotrophin-releasing hormone agonist during the luteal phase in IVF. Hum Reprod. 2001 Aug;16(8):1671-5. doi: 10.1093/humrep/16.8.1671. PMID 11473961
- [Result] Isik AZ, Caglar GS, Sozen E, Akarsu C, Tuncay G, Ozbicer T, Vicdan K. Single-dose GnRH agonist administration in the luteal phase of GnRH antagonist cycles: a prospective randomized study. Reprod Biomed Online. 2009 Oct;19(4):472-7. doi: 10.1016/j.rbmo.2009.04.001. PMID 19909586
- [Result] Bar Hava I, Blueshtein M, Ganer Herman H, Omer Y, Ben David G. Gonadotropin-releasing hormone analogue as sole luteal support in antagonist-based assisted reproductive technology cycles. Fertil Steril. 2017 Jan;107(1):130-135.e1. doi: 10.1016/j.fertnstert.2016.10.011. Epub 2016 Oct 27. PMID 28228316
- [Result] Aboulghar MA, Marie H, Amin YM, Aboulghar MM, Nasr A, Serour GI, Mansour RT. GnRH agonist plus vaginal progesterone for luteal phase support in ICSI cycles: a randomized study. Reprod Biomed Online. 2015 Jan;30(1):52-6. doi: 10.1016/j.rbmo.2014.09.017. Epub 2014 Oct 13. PMID 25456166
- [Result] Chen SL, Wu FR, Luo C, Chen X, Shi XY, Zheng HY, Ni YP. Combined analysis of endometrial thickness and pattern in predicting outcome of in vitro fertilization and embryo transfer: a retrospective cohort study. Reprod Biol Endocrinol. 2010 Mar 24;8:30. doi: 10.1186/1477-7827-8-30. PMID 20334664
- [Result] Ye H, Luo X, Pei L, Li F, Li C, Chen Y, Zhang X, Huang G. The addition of single dose GnRH agonist to luteal phase support in artificial cycle frozen embryo transfer: a randomized clinical trial. Gynecol Endocrinol. 2019 Jul;35(7):618-622. doi: 10.1080/09513590.2018.1563888. Epub 2019 Jan 31. PMID 30700175